CLINICAL TRIAL: NCT04119635
Title: Treatment and Long-term Outcomes of Pediatric Patient With Penetrating Crohn's Disease: the Multicenter Cross-sectional Study
Brief Title: Pediatric Penetrating Crohn's Disease
Acronym: Pediatric B3
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Pediatric gastroenterology service, Toulouse University Hospital: Dr Breton (Unknown); Adult gastroenterology service, Montpellier University Hospital: Dr Pineton de Chambrun (Unknown); Pediatric gastroenterology service, Montpellier University Hospital: Dr Kollen (Unknown); EPIMAD Registry: Dr Gower-Rousseau (Unknown)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0366
Record Dates: First submitted 2019-10-02; First posted 2019-10-08 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Pediatric Penetrating Crohn's Disease
Keywords: Crohn's disease; Penetrating complication; Pediatric; Inflammatory bowel disease
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The incidence of Crohn's disease (CD) increased the last few years, especially in children, with 20% percent of CD patients diagnosed during childhood. The CD is a chronic disease without curative treatment, medical or surgical, and evolution is longer in children, avoid iterative digestive resections and their consequences in these patients is a major issue.

The beginning of the disease at pediatric age is considered to be a poor prognostic factor and is considered to be more aggressive than that of adults: more extensive, more active and requiring more immunosuppressive treatments, with a more frequent dependence on corticosteroids and a shorter delay between the beginning of symptoms and the first surgery. After 5 years of evolution, 13 to 50% of patients with early pediatric MC have undergone intestinal resection.

The Paris' classification defined 3 phenotypes or behaviors in pediatric Crohn's disease. Penetrating phenotype (B3) is a heterogeneous group defined by the presence of intra-abdominal perforation, fistulas or abscesses. The B3 phenotype is a risk factor for pejorative evolution in CD with a risk increased of surgical resection.

In the pediatric population, the natural history of patients with penetrating CD is unknown. Most studies focus on CD beginning at pediatric age but with penetrating complications occurring in adulthood or pediatric penetrating CD but with relatively short follow-up. The risk of recurrence of the penetrating disease after a first complication in childhood is unknown, the factors influencing this risk also. And, there is no consensus either concerning optimal B3 management in children, and the practices are variable from specialist to specialist.

After describing the pediatric population with penetrating CD, the aim of this study was to know the incidence of bowel resection for B3 episode. The secondary aims were to describe the immediate management and long-term evolution of these patients and to identify risk factors for adverse evolution.

DETAILED DESCRIPTION:
This study is cross-sectional and is carrying out between 1995 and 2017 in two French tertiary referral centers (Montpellier, Toulouse) and EPIMAD registry which is currently the largest Inflammatory Bowel Disease cohort in world and cover 9.6% of French population (Nord, Pas-de-Calais, Somme, and Seine-Maritime department).

All patients diagnosed with CD who had underwent a B3 complication (intra-abdominal abscess, fistula, perforation, peritonitis, or phlegmon) before the age of 18. Patient having isolated perineal disease, indeterminate colitis or with too much missing data were excluded.

The main endpoint: incidence of intestinal resection performed for B3 complication.

The secondary endpoints:

* description of the pediatric population with B3 complication with:
* demographic data: sex, family history, phenotype of the disease according to the Paris classification, age at diagnosis of B3, period of diagnosis of B3 (before or after 2001), time between the diagnosis of CD and the diagnosis of B3, a history of medical and surgical treatment for CD received before B3.
* clinical data: type of B3 complication, presence of stenosis and its location, clinical symptoms (fever, obstructive symptoms), nutritional status.
* description of the immediate management of these patients, specifying: the place of care, the type of immediate management performed, the drug treatments received in the acute phase, the medical treatments for CD introduced for the B3 episode, the intestinal resections performed for the B3 episode, the realization of a stoma, the radiological drainage of abscesses, the immediate complications of B3.
* description of the long-term evolution of these patients, specifying: the given drug treatments, the clinical recurrence of the CD, the recurrence of B3, the need for intestinal resection during follow-up, the occurrence of other events
* identification of risk factors for pejorative evolution defined by "recurrence of B3" or "intestinal resection" in these patients.

ELIGIBILITY:
Inclusion criteria:

- patients diagnosed with CD who had underwent a B3 complication (intra-abdominal abscess, fistula, perforation, peritonitis, or phlegmon)

Exclusion criteria:

* patient having isolated perineal disease, indeterminate colitis or with too much missing data were excluded
* patients refuse the use of medical data will be excluded.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients diagnosed with CD who had underwent a B3 complication (intra-abdominal abscess, fistula, perforation, peritonitis, or phlegmon) before the age of 18
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
incidence of intestinal resection performed for B3 complication in pediatric population | through study completion, an average of 10 years
  * Incidence of intestinal resection at the first episode of B3
  * Cumulated incidence of intestinal resection in the follow up.

SECONDARY OUTCOMES:
incidence of recurrence of B3 complication in pediatric population | through study completion, an average of 10 years
  Incidence of recurrence of B3 complication and specifying :
  * median duration of recurrence after the first episode
  * number of recurrence
identification of risk factors for pejorative evolution (recurrence of <B3 or intestinal resection) of the pediatric population with B3 complication | through study completion, an average of 10 years.
  Multivariate analysis with the following data to define parameters associated with "recurrence of B3" or "intestinal resection"

CONTACTS AND LOCATIONS:
Overall Officials: Laura Kollen, MD, Principal Investigator — University Hospitals of Montpellier
Locations (1):
- Uh Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC